CLINICAL TRIAL: NCT05787977
Title: The Effect of Treadmill Training With Visual Feedback and Rhythmic Auditory Cue on Gait and Balance in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Asma001-04
Record Dates: First submitted 2023-02-20; First posted 2023-03-28 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Treadmill training; Visual Feedback and Rhythmic Auditory cue; Gait and Balance; Hemiplegic Cerebral palsy
MeSH Terms: interventions — Feedback, Sensory

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Treadmil Training with visual feedback and rhythmic Auditory Cue
  Interventions: Other: Visual Feedback and Rhythmic Auditory Cue
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Other: Visual Feedback and Rhythmic Auditory Cue — Patients were trained five times per week for eight weeks. After eight weeks of training the gait pattern and balance was evaluated by the gait parameters, 6min Walk test, Pediatric Balance Scale and Berg balance scale.
  Arms: Interventional Group

SUMMARY:
The development of efficient and independent walking is an important therapeutic goal for many children with cerebral palsy (CP). Consequently, there has been growing interest in determining the effects of treadmill training programs for these children.

This study helped to investigates the effect of treadmill training with visual feedback and rhythmic auditory cue (VF+RAC) for walking symmetry and balance ability. Participants were chosen from Sehat medical complex and they were randomly allocated to either the VF+RAC or the Control group. The VF+RAC group received treadmill training with VF and RAC, and the Control group undergo treadmill training without any visual and auditory stimulation. VF+RAC and Control groups was trained five times per week for eight weeks. After eight weeks of training the gait pattern and balance were evaluated by the gait parameters, 6min Walk test, Pediatric Balance Scale and Berg balance scale.

DETAILED DESCRIPTION:
Cerebral palsy is the most common cause of childhood-onset, lifelong physical disability in most countries, affecting about 1 in 500 neonates with an estimated prevalence of 17 million people worldwide. Cerebral palsy is a non-progressive brain injury or lesion acquired during the antenatal, perinatal or early postnatal period. The clinical manifestations of cerebral palsy vary greatly in the type of movement disorder, the degree of functional ability and limitation and the affected parts of the body.

Auditory entrainment can influence gait performance in movement disorders. The entrainment can incite neurophysiological and musculoskeletal changes to enhance motor execution. Biofeedback systems have been extensively used in walking exercises for gait improvement.

ELIGIBILITY:
Inclusion Criteria:

* children having GMF level 1 and 2,
* willing to participate,
* Pediatric subjects Diagnosed with cerebral palsy, receiving Neurodevelopmental
* Rehabilitation program regularly.

Exclusion Criteria

* Child using any sort of auditory aid
* Children with visual limitation,
* Child using orthosis for lower extremity

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
6 Minutes Walk Test | Change from baseline at 8th week
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Pediatric Balance scale | Change from baseline at 8th Week
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
Berg Balance Scale | Change from baseline at 8th week
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.

CONTACTS AND LOCATIONS:
Overall Officials: Momina Mehmood, Principal Investigator — University of Lahore
Locations (1):
- Sehat Medical Complex, Lahore, Lahore, Punjab Province, Pakistan